CLINICAL TRIAL: NCT05537454
Title: Maternal Stress, Human Milk Composition, and Neurodevelopmental and Feeding Outcomes
Brief Title: Maternal Stress, Milk Composition, and Preterm Neurodevelopment
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: SPH-2022-31233
Record Dates: First submitted 2022-09-01; First posted 2022-09-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explores the associations between maternal stress, breastmilk composition, and feeding and neurodevelopment for preterm infants in the NICU and at 4 months corrected age.

DETAILED DESCRIPTION:
The proposed study will address our novel hypothesis that maternal stress is associated with feeding outcomes and markers of impaired neurodevelopment for preterm infants and alters human milk and infant gut profiles in ways that affect preterm neurodevelopment.

Mothers and their preterm infants (28-34 weeks gestation at birth) will be recruited to determine if: (1) variation in postnatal stress among mothers of very preterm infants relates to the total volume or proportion of maternal milk provided to her infant in the NICU and if (2) variation in maternal postnatal stress relates to her preterm infant's neurocognitive status at NICU discharge and 4 months corrected age. This project also involves collection/storage of maternal milk and infant fecal samples for multi-omics analyses. More specifically, the study will address: (3A) Is maternal postnatal stress associated with the metabolomic and microbiome characteristics of the infant's gut and/or the milk composition?, and (3B) Do milk composition differences relate to infant neurodevelopment? The aims of the proposed study contribute to our overarching research goal, which is to improve neurodevelopmental health for preterm infants by building the health and resilience of the mother-milk-infant triad.

ELIGIBILITY:
Inclusion Criteria:

* preterm infant born between 28 0/7 and 34 6/7 weeks' gestation that are medically stable for study procedures
* mother of preterm infant meeting criteria and a) 18 to 45 years of age at the time of delivery

Exclusion Criteria:

* infants: major congenital anomalies, anticipated death, positive blood culture at birth, hypoxic ischemic encephalopathy, grade IV intraventricular hemorrhage, or plan to transfer care before discharge (35-37 weeks postmenstrual age).
* mothers: a) alcohol consumption >1 drink per week or any tobacco consumption during pregnancy, b) known congenital metabolic, endocrine disease or congenital illness affecting infant feeding/growth

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Early preterm infants and their mothers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Maternal milk production inpatient | 28-35 weeks postmenstrual age
  total volume (mL)
Maternal milk production 4 months corrected age | 4 months corrected age
  total volume (mL)
Maternal milk proportion inpatient | 28-35 weeks postmenstrual age
  Proportion of maternal milk vs donor milk/formula (%)
Maternal milk proportion 4 months corrected age | 4 months corrected age
  Proportion of maternal milk vs donor milk/formula (%)
Infant Neurodevelopment inpatient | 35-37 weeks postmenstrual age
  event related potentials (ERP)
Infant Neurodevelopment 4 months corrected age | 4 months corrected age
  event related potentials (ERP)
Infant Neurodevelopment 4 months corrected age | 4 months corrected age
  visual evoked potentials (VEP)
Infant gut microbiome inpatient | 28-35 weeks postmenstrual age
  Microbial diversity of fecal samples
Infant gut microbiome 4 months corrected age | 4 months corrected age
  Microbial diversity of fecal samples
Milk microbiome inpatient | 28-35 weeks postmenstrual age
  Microbial diversity of milk samples
Milk microbiome 4 months corrected age | 4 months corrected age
  Microbial diversity of milk samples
Milk metabolome inpatient | 28-35 weeks postmenstrual age
  Concentration of untargeted and targeted metabolites
Milk metabolome 4 months corrected age | 4 months corrected gestational age
  Concentration of untargeted and targeted metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data upon request
Time Frame: Data will be made available to other researchers no later than the acceptance for publication of the main findings from the final dataset. Depending on the volume of data requests from external researchers, a long term data sharing and preservation plan may be used to store and make publicly accessible the data beyond the life of the project.